CLINICAL TRIAL: NCT00978549
Title: Randomised Phase III Study of Docetaxel vs Active Symptom Control in Patients With Relapsed Oesophago-gastric Adenocarcinoma
Brief Title: Symptom Control With or Without Docetaxel in Treating Patients With Relapsed Esophageal Cancer or Stomach Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CRCA-COUGAR-02; CDR0000649670 (Registry Identifier: PDQ (Physician Data Query)); EudraCT-2006-005046-37; ISRCTN13366390; CRUK/07/013; EU-20969
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2009-09

CONDITIONS: Adenocarcinoma of the Gastroesophageal Junction; Esophageal Cancer; Gastric Cancer; Nausea and Vomiting; Pain
Keywords: pain; nausea and vomiting; adenocarcinoma of the esophagus; adenocarcinoma of the stomach; adenocarcinoma of the gastroesophageal junction; recurrent gastric cancer; stage IIIA gastric cancer; stage IIIB gastric cancer; stage IIIC gastric cancer; stage IV gastric cancer; recurrent esophageal cancer; stage IIIA esophageal cancer; stage IIIB esophageal cancer; stage IIIC esophageal cancer; stage IV esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Nausea; Vomiting; Pain; Adenocarcinoma Of Esophagus | interventions — Docetaxel; Analgesia; Radiotherapy

INTERVENTIONS:
Drug: docetaxel
Drug: steroid therapy
Other: questionnaire administration
Procedure: nausea and vomiting therapy
Procedure: pain therapy
Procedure: quality-of-life assessment
Procedure: standard follow-up care
Radiation: radiation therapy

SUMMARY:
RATIONALE: Analgesics, antiemetics, steroids, and radiation therapy are effective in helping to control symptoms caused by cancer. It is not yet known whether these treatments are more effective when given with or without docetaxel in treating patients with relapsed esophageal cancer or stomach cancer.

PURPOSE: This randomized phase II trial is studying symptom control given together with docetaxel to see how well it works compared with symptom control given without docetaxel in treating patients with relapsed esophageal cancer or stomach cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare overall survival of patients with relapsed adenocarcinoma of the esophagus or stomach after treatment with docetaxel and active symptom control vs active symptom control alone.

Secondary

* To determine the time to documented progression in patients treated with docetaxel.
* To assess response rates to docetaxel in patients treated with docetaxel.
* To determine toxicity of docetaxel in patients treated with docetaxel.
* To assess the quality of life of these patients.
* To evaluate the health economic impact.

OUTLINE: This is a multicenter study.

Patients are stratified according to stage (locally advanced vs metastatic), site of disease (esophagus vs esophagogastric junction vs stomach), duration of response to prior chemotherapy (no response vs response duration < 3 months vs response duration 3-6 months), and ECOG performance status (0-1 vs 2). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive docetaxel IV over 1 hour on day 1 and active symptom control (e.g., analgesics [including opioids], antiemetics, steroids, palliative radiotherapy) daily.
* Arm II: Patients receive active symptom control as in arm I. Courses repeat every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients in arm I undergo tissue biopsy collection at baseline and after 3 courses of treatment for biomarker analysis.

Quality of life is assessed by the QLQ-C30 and QLQ-STO22 questionnaires at baseline and at 3, 6, 9, 12, 18, and 24 weeks. Health resource use is assessed by the EQ-5D questionnaire at baseline and then periodically during and after treatment.

After completion of study treatment, patients are followed up every 6 weeks for 1 year and then every 3 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the esophagus or stomach, including adenocarcinoma of the esophagogastric junction

  * Advanced disease not amenable to curative treatment
  * Documented progressive disease while receiving or within 6 months of completion of first-line chemotherapy with a platinum- and fluoropyrimidine-based therapy either for advanced disease or as neoadjuvant/perioperative therapy
* No cerebral or leptomeningeal metastasis

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* Hemoglobin ≥ 10 g/dL
* WBC ≥ 3.0 x 10^9/L
* ANC ≥ 1.5 x 10^9/L
* Platelets ≥ 100 x 10^9/L
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Total bilirubin normal
* ALT ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 3 months after completion of treatment
* No clinically significant peripheral neuropathy (grade 2-4)
* No prior malignancy except for curatively treated basal cell carcinoma of the skin or cervical intraepithelial neoplasia
* No medical or psychiatric condition that would influence the ability of patients to provide informed consent
* No other serious or uncontrolled illness that, in the opinion of the investigator, makes it undesirable for the patient to enter the trial

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy with taxanes

  * ≤ 1 prior chemotherapy regimen in advanced setting allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-04 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Time to documented progression (arm I)
Response rate (arm I)
Toxicity (arm I)
Quality of life as assessed by EORTC QLQ-C30 and -STO22
Health economic evaluation as assessed by EQ-5D

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Ford, MD, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (8):
- United Kingdom (8):
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Warwick Medical School Clinical Trials Unit, Coventry, England
  - St. Luke's Cancer Centre at Royal Surrey County Hospital, Guildford, England
  - Medical Research Council Clinical Trials Unit, London, England
  - Royal South Hants Hospital, Southampton, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales